CLINICAL TRIAL: NCT01298440
Title: The Effect of Intravitreal Bevacizumab (Avastin) Injection on Retinal Blood-Flow Velocity in Patients With Choroidal Neovascularization
Brief Title: Bevacizumab Effect on Blood Velocity
Status: Completed | Type: Observational
Sponsor: Optical Imaging, Ltd. (Industry)
Responsible Party: Optical Imaging, Ltd
Other Study IDs: AvastinRFI
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Choroidal Neovascularization
MeSH Terms: conditions — Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Retinal blood flow velocity is affected by Bevacizump intravitreal injection. This effect is correlated to treatment success.

DETAILED DESCRIPTION:
The purpose of the study was to carry out a pilot study on the short-term effect of intravitreal Bevacizumab (Avastin) injection on retinal blood-flow velocity and test whether the short-term haemodynamic changes could predict the longer term clinical result of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CNV receiving Bevacizumab intravitreal injection

Exclusion Criteria:

* Candidates in whom the retina could not be seen clearly because of media opacity or a poorly dilating pupil

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with choroidal neovascularization (CNV)
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Blood flow velocity change | 1 day following injection

CONTACTS AND LOCATIONS:
Overall Officials: Adiel Barak, MD, Principal Investigator — Tel aviv university Sackler school of medicine
Locations (1):
- Tel aviv sourasky medical center, Tel Aviv, Israel

REFERENCES:
- [Derived] Burgansky-Eliash Z, Lowenstein A, Neuderfer M, Kesler A, Barash H, Nelson DA, Grinvald A, Barak A. The correlation between retinal blood flow velocity measured by the retinal function imager and various physiological parameters. Ophthalmic Surg Lasers Imaging Retina. 2013 Jan-Feb;44(1):51-8. doi: 10.3928/23258160-20121221-13. PMID 23418734